CLINICAL TRIAL: NCT02213146
Title: A Double-blinded, Randomised, Three-period Crossover Euglycaemic Clamp Trial Investigating the Pharmacokinetics, Glucodynamics and Safety of BioChaperone Human Insulin, Human Insulin (Huminsulin® Normal) and Insulin Lispro (Humalog®) in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BC3-CT010
Record Dates: First submitted 2014-08-08; First posted 2014-08-11 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2015-06

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BioChaperone human insulin (Experimental): BioChaperone Human Insulin
  Interventions: Drug: BioChaperone human insulin; Drug: Huminsulin® Normal; Drug: Humalog®
- Human insulin (Active Comparator): Huminsulin® Normal
  Interventions: Drug: BioChaperone human insulin; Drug: Huminsulin® Normal; Drug: Humalog®
- Insulin lispro (Active Comparator): Humalog®
  Interventions: Drug: BioChaperone human insulin; Drug: Huminsulin® Normal; Drug: Humalog®

INTERVENTIONS:
Drug: BioChaperone human insulin — Single dose of 0.2 U/kg body weight injected subcutaneously
Drug: Huminsulin® Normal — Single dose of 0.2 U/kg body weight injected subcutaneously
Drug: Humalog® — Single dose of 0.2 U/kg body weight injected subcutaneously

SUMMARY:
The addition of BioChaperone to already marketed prandial human insulin preparations may accelerate the onset and shorten the duration of action due to facilitation of the insulin absorption after subcutaneous injection.

The aim of the trial is to assess the efficacy and safety of BioChaperone human insulin in subjects with type 1 diabetes under a dose of 0.2 U/kg.

This trial is a single center, randomised, double-blinded, three treatment, three-period cross-over, 10-hour euglycaemic clamp trial in subject with type 1 diabetes mellitus. Each subject will be randomly allocated to a single dose of BioChaperone human insulin 0.2 U/kg, a single dose of Huminsulin® Normal 0.2 U/kg and a single dose of Humalog® 0.2 U/kg on 3 separate dosing visits.

ELIGIBILITY:
Inclusion Criteria:

* Male subject with type 1 diabetes for at least 12 months
* Treated with multiple daily insulin injections or insulin pump (CSII) for at least 12 months
* Body mass index: 18.5-28.0 kg BW·m-2
* HbA1c: ≤ 9.0%

Exclusion Criteria:

* Diabetes mellitus type 2
* Receipt of any investigational product within 3 months prior to first dosing of investigational product in this trial
* Clinically significant abnormalities as judged by the Investigator
* Any systemic treatment with drugs known to interfere with glucose metabolism
* History of alcoholism or drug/chemical abuse as per Investigator's judgement
* Use of any tobacco or nicotine-contained product within one year prior to screening

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUCins(0-1h)) | 1 hour
  Area under the human insulin serum concentration - time curve from t=0 to 1 hour

SECONDARY OUTCOMES:
Pharmacokinetics: Early t0.5max ins/lisp | up to 10 hours post administration
  Time to first observed half maximum serum human insulin / insulin lispro concentration
Glucodynamics: Area under the glucose infusion rate - time curve from t=0 to 10 hours | 10 hours
  Area under the glucose infusion rate - time curve from t=0 to 10 hours
Glucodynamics: Early t0.5 Glucose Infusion Rate max (GIRmax) | 10 hours
  Time to first observed half maximum glucose infusion rate
Glucodynamics: GIRmax - Maximum glucose infusion rate | 10 hours
  Maximum glucose infusion rate
Pharmacokinetics: AUCins/lisp(0-10h): Area under the human insulin / insulin lispro serum concentration | 10 hours
  Area under the human insulin / insulin lispro serum concentration - Time curve from t=0 to 10 hours
Pharmacokinetics: Tmax(ins/lisp) - Time to maximum observed serum human insulin concentration and insulin lispro concentration | 10 hours
  Time to maximum observed serum human insulin concentration and insulin lispro concentration
Safety and tolerability: adverse events, local tolerability, vital signs variation, ECG, laboratory safety parameters | up to 7 weeks
  Adverse events, local tolerability, vital signs variation, ECG, laboratory safety parameters
Pharmacokinetics: Cmax(ins/lisp) | up to 10 hours
  Maximum observed human insulin / insulin lispro serum concentration
Glucodynamics: Area under the glucose infusion rate - time curve from t=0 to 2 hours | 2 hours post administration
  Area under the glucose infusion rate - time curve from t=0 to 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Grit Andersen, MD, Principal Investigator — Profil GmbH
Locations (1):
- Profil GmbH, Neuss, Germany